CLINICAL TRIAL: NCT05222607
Title: LONG RUN: LONGitudinal Evaluation and Real-world Evidence of Uniquely Purified incobotulinumtoxinA (Xeomin) in Treatment Naïve Participants
Brief Title: Longitudinal Evaluation and Real-world Evidence of NT201
Status: Terminated | Type: Observational
Why Stopped: Corporate Management Decision
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: M602011076
Record Dates: First submitted 2021-12-23; First posted 2022-02-03 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Glabellar Frown Lines and Canthal Lines and/or Horizontal Forehead Lines in the Upper Face
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Facial treatment with incobotulinumtoxinA in treatment naïve participants
  Interventions: Drug: IncobotulinumtoxinA

INTERVENTIONS:
Drug: IncobotulinumtoxinA — IncobotulinumtoxinA injections for aesthetic indications.
  Other Names: XEOMIN®; BOCOUTURE®

SUMMARY:
This study is to collect long-term real-world evidence data from clinics in several countries in order to obtain an improved understanding of the safety and effectiveness of incobotulinumtoxinA in botulinum neurotoxin type A (BoNT-A) treatment naïve participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Planning treatment with incobotulinumtoxinA.

Exclusion Criteria:

* Any contraindication to treatment with incobotulinumtoxinA or any other neurotoxins.
* Currently pregnant, breastfeeding, or intending to become pregnant during study participation.
* Known hypersensitivity to incobotulinumtoxinA or any of its formulation ingredients.
* Any infection and/or inflammation at the planned injection points.
* Previous treatment with any botulinum toxin products for any aesthetic or therapeutic indications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants, 18 years of age or older, seeking treatment with incobotulinumtoxinA for UFL in the North American, Latin American, European, and Asia-Pacific regions.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Assessment of FACE-Q Patient-Perceived Age Visual Analogue Scale mean change | Up to 3 years
  Explore the effectiveness of the incobotulinumtoxinA injections in treatment naïve participants for facial cosmetic procedures during up to 3 years continuous treatment exposure, as measured by assessment of FACE-Q Patient-Perceived Age Visual Analogue Scale mean change from first treatment visit to the 4-to-6 weeks timepoint.

SECONDARY OUTCOMES:
Assessment of FACE-Q Satisfaction with Decision Scale mean change | Up to 3 years
  Explore the effectiveness of the incobotulinumtoxinA injections in treatment naïve participants for facial cosmetic procedures during up to 3 years continuous treatment exposure, as measured by assessment of FACE-Q Satisfaction with Decision Scale mean change from first treatment visit to the 4-to-6 weeks timepoint.

CONTACTS AND LOCATIONS:
Locations (1):
- SkinDC, Arlington, Virginia, United States